CLINICAL TRIAL: NCT01916967
Title: A Phase III Multicentre, Parallel-group, Randomized, Placebo-controlled, Double-blind Clinical Trial to Study the Efficacy and Safety of MK-4117 in Japanese Subjects With Chronic Urticaria.
Brief Title: An Efficacy and Safety Study of Desloratadine (MK-4117) in Japanese Participants With Chronic Urticaria (MK-4117-201)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4117-201; 132243 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2013-08-02; First posted 2013-08-06 (Estimated); Results first posted 2014-10-30 (Estimated); Last update posted 2024-06-18 (Actual); Status verified 2022-02

CONDITIONS: Urticaria
Keywords: Urticaria; Skin Diseases, Vascular; Skin Diseases; Hypersensitivity, Immediate; Hypersensitivity; Immune System Diseases; Cholinergic Antagonists; Cholinergic Agents; Neurotransmitter Agents; Histamine H1 Antagonists, Non-Sedating; Histamine H1 Antagonists; Histamine Antagonists; Histamine Agents
MeSH Terms: conditions — Urticaria; Skin Diseases, Vascular; Skin Diseases; Hypersensitivity, Immediate; Hypersensitivity; Immune System Diseases | interventions — desloratadine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Desloratadine 5 mg (Experimental): Participants receive desloratadine 5 mg, as one 5-mg tablet and one placebo tablet, orally, once daily in the evening for 2 weeks
  Interventions: Drug: Desloratadine; Drug: Placebo
- Desloratadine 10 mg (Experimental): Participants receive desloratadine 10 mg, as two 5-mg tablets, orally, once daily in the evening for 2 weeks
  Interventions: Drug: Desloratadine
- Placebo (Placebo Comparator): Participants receive placebo, as two tablets, orally, once daily in the evening for 2 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Desloratadine — Desloratadine 5 mg tablets, given orally, once daily in the evening for 2 weeks
  Arms: Desloratadine 10 mg; Desloratadine 5 mg
Drug: Placebo — Placebo tablets, given orally, once daily in the evening for 2 weeks
  Arms: Desloratadine 5 mg; Placebo

SUMMARY:
This is a study to evaluate the efficacy and safety of desloratadine (MK-4117) in Japanese participants with chronic urticaria. The primary hypothesis is that the efficacy of desloratadine 10 mg and 5 mg is superior to placebo as based on the change from Baseline in the sum score of pruritus/itch and rash as assessed by the Investigator at Week 2.

ELIGIBILITY:
Inclusion Criteria:

* Chronic urticaria [rash (erythema, wheal) for more than 1 month without any known cause]
* Out-patient

Exclusion Criteria:

* Stimulation-induced urticaria [physical urticaria (e.g. cold, solar, and heat urticaria), cholinergic urticaria, contact urticaria)]
* Hypersensitivity to antihistamines or ingredients of a study drug

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2013-08-27 (Actual); Primary Completion 2014-02-28 (Actual); Study Completion 2014-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hide M, Maeda Y, Oshima N, Hisada S. A Phase III clinical trial of desloratadine in Japanese subjects with chronic urticaria: A randomized controlled trial. J Clin Therapeut Med. 2016;32(11):891-903.. [in Japanese] https://mol.medicalonline.jp/archive/search?jo=an9cltmd&ye=2016&vo=32&issue=11

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Desloratadine 5 mg | Desloratadine 10 mg | Placebo
Started | 80 | 79 | 80
Completed | 80 | 78 | 71
Not Completed | 0 | 1 | 9
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Lack of Efficacy | 0 | 0 | 6
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Desloratadine 5 mg | Desloratadine 10 mg | Placebo | Total
Number analyzed (Participants) | 80 | 79 | 80 | 239
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.4 (16.3) | 40.6 (15.8) | 39.3 (15.2) | 39.4 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 48 | 45 | 152
  Male | 21 | 31 | 35 | 87

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Sum Score of Pruritus/Itch and Rash Assessed by Investigator at Week 2
Description: The Investigator assessed the severity of participant pruritus/itch during the daytime (0=Virtually no itching to 4=Cannot relax because of constant itching) and nighttime (0=Virtually no itching to 4=Cannot sleep because of itching). The score used for pruritus/itch was the higher of the day or night scores (0=Asymptomatic to 4=Severe). The Investigator also assessed the severity of participant rash using the overall rash score (0=No rash to 3=Looks very bad). The sum of the pruritus/itch score (0-4) and rash score (0-3) could range from 0 to 7, with a higher sum score indicating greater severity. The change from Baseline in the sum of the pruritus/itch and overall rash scores at the Week 2 clinic visit was calculated.
Time Frame: Baseline Visit and Week 2 Visit
Population: The Full Analysis Set (FAS) population consisted of all randomized participants who took at least one dose of study drug, had a Baseline assessment and a Week 2 assessment for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Desloratadine 5 mg | Desloratadine 10 mg | Placebo
Number analyzed (Participants) | 80 | 79 | 80
Score on a Scale | -3.19 [-3.56 to -2.83] | -3.16 [-3.52 to -2.79] | -2.02 [-2.40 to -1.65]
Statistical Analysis 1: Comparison: Desloratadine 5 mg vs Placebo; Difference in least squares (LS) means of Desloratadine 5 mg and Placebo; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis; Model with terms of visit, visit-by-treatment, visit-by-age strata, visit-by-severity interactions; visit treated as a categorical variable; Difference in LS means = -1.17, 95% CI 2-sided [-1.69 to -0.65]
Statistical Analysis 2: Comparison: Desloratadine 10 mg vs Placebo; Difference in LS means of Desloratadine 10 mg and Placebo; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LS means = -1.13, 95% CI 2-sided [-1.66 to -0.61]

2. Primary Outcome: Number of Participants Who Experienced at Least One Adverse Event (AE)
Description: An AE is any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study drug or protocol-specified procedure, whether or not considered related to the study drug or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of the study drug, is also an AE.
Time Frame: Up to 4 weeks (Up to 2 weeks after last dose of study drug)
Population: The Safety Population consisted of all participants who received at least one dose of study drug. One Placebo group participant took the wrong study drug. This participant was analyzed separately.
Measure: Number; unit: Participants
Groups:
- Desloratadine 5 mg→Placebo: Participant received desloratadine 5 mg, as one 5-mg tabet and one placebo tablet, orally, once daily for 1 week and then received placebo, as two tablets, orally, once daily for 1 week
Arm/Group | Desloratadine 5 mg | Desloratadine 10 mg | Placebo | Desloratadine 5 mg→Placebo
Number analyzed (Participants) | 80 | 79 | 79 | 1
Participants | 24 | 18 | 16 | 0

3. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an AE
Description: as for outcome 2
Time Frame: Up to 2 weeks
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Desloratadine 5 mg | Desloratadine 10 mg | Placebo | Desloratadine 5 mg→Placebo
Number analyzed (Participants) | 80 | 79 | 79 | 1
Participants | 0 | 0 | 2 | 0

4. Secondary Outcome: Change From Baseline in the Sum Score of Pruritus/Itch and Rash Assessed by Investigator at Day 3 and Week 1
Description: The Investigator assessed the severity of participant pruritus/itch during the daytime (0=Virtually no itching to 4=Cannot relax because of constant itching) and nighttime (0=Virtually no itching to 4=Cannot sleep because of itching). The score used for pruritus/itch was the higher of the day or night scores (0=Asymptomatic to 4=Severe). The Investigator also assessed the severity of participant rash using the overall rash score (0=No rash to 3=Looks very bad). The sum of the pruritus/itch score (0-4) and rash score (0-3) could range from 0 to 7, with a higher sum score indicating greater severity. The changes from Baseline in the sum of the pruritus/itch and overall rash scores at the Day 3 and Week 1 clinic visits were calculated.
Time Frame: Baseline Visit and Day 3 Visit, Week 1 Visit
Population: The FAS population consisted of all randomized participants who took at least one dose of study drug, had a Baseline assessment and at least one post-Baseline assessment for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Desloratadine 5 mg | Desloratadine 10 mg | Placebo
Number analyzed (Participants) | 80 | 79 | 80
Score on a Scale
  Change from Baseline at Day 3 | -2.57 [-2.91 to -2.23] | -2.75 [-3.09 to -2.41] | -0.80 [-1.14 to -0.46]
  Change from Baseline at Week 1 | -3.01 [-3.34 to -2.68] | -3.16 [-3.50 to -2.83] | -1.39 [-1.72 to -1.06]

5. Secondary Outcome: Change From Baseline in the Pruritus/Itch Score Assessed by Investigator at Day 3, Week 1 and Week 2
Description: The Investigator assessed the severity of participant pruritus/itch during the daytime and nighttime (0=Asymptomatic to 4=Severe). The sum of the daytime and nighttime pruritus/itch scores could range from 0 to 8, with a higher score indicating greater severity. The changes from Baseline in the sum of the daytime and nighttime scores at the Day 3, Week 1 and Week 2 clinic visits were calculated.
Time Frame: Baseline Visit and Day 3 Visit, Week 1 Visit, Week 2 Visit
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Desloratadine 5 mg | Desloratadine 10 mg | Placebo
Number analyzed (Participants) | 80 | 79 | 80
Score on a Scale
  Change from Baseline at Day 3 | -2.62 [-2.97 to -2.27] | -2.72 [-3.07 to -2.37] | -0.61 [-0.95 to -0.26]
  Change from Baseline at Week 1 | -2.98 [-3.35 to -2.61] | -3.13 [-3.50 to -2.76] | -1.38 [-1.75 to -1.01]
  Change from Baseline at Week 2 | -3.17 [-3.56 to -2.77] | -3.21 [-3.60 to -2.81] | -1.91 [-2.31 to -1.50]

6. Secondary Outcome: Change From Baseline in the Rash Score Assessed by Investigator at Day 3, Week 1 and Week 2
Description: The Investigator assessed the severity of participant rash (erythema: 0=no symptom to 3=intensive redness, and wheal: 0=no symptom to 3=significant ridge). The sum score for erythema plus wheal could range from 0 to 6, with a higher score indicating greater severity. The changes from Baseline in the sum score for erythema plus wheal at the Day 3, Week 1 and Week 2 clinic visits were calculated.
Time Frame: Baseline Visit and Day 3 Visit, Week 1 Visit, Week 2 Visit
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Desloratadine 5 mg | Desloratadine 10 mg | Placebo
Number analyzed (Participants) | 80 | 79 | 80
Score on a Scale
  Change from Baseline at Day 3 | -2.31 [-2.63 to -2.00] | -2.61 [-2.93 to -2.29] | -0.99 [-1.31 to -0.67]
  Change from Baseline at Week 1 | -2.65 [-2.97 to -2.33] | -2.98 [-3.30 to -2.66] | -1.44 [-1.76 to -1.12]
  Change from Baseline at Week 2 | -2.94 [-3.28 to -2.61] | -2.91 [-3.25 to -2.57] | -1.98 [-2.33 to -1.64]

7. Secondary Outcome: Number of Participants With a Moderate or Remarkable Improvement in the Global Improvement Rate of Both Pruritus/Itch and Rash (Erythema and Wheal) Assessed by the Investigator at Day 3, Week 1 and Week 2
Description: The global improvement judgment criteria were used to assess overall improvement in pruritus/itch and rash. The Investigator assessed participant global improvement according to 5 grades (Grade 1=Remarkable improvement to Grade 5=Aggravated). The number of participants with moderate or remarkable improvements was calculated. Remarkable improvement (Grade 1) was defined as both pruritus/itch and rash (erythema and wheal) disappeared, or pruritus/itch disappeared and rash (erythema and wheal) was apparently improved. Moderate improvement (Grade 2) was defined as both pruritus/itch and rash (erythema and wheal) were greatly improved.
Time Frame: Baseline Visit and Day 3 Visit, Week 1 Visit, Week 2 Visit
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Desloratadine 5 mg | Desloratadine 10 mg | Placebo
Number analyzed (Participants) | 80 | 79 | 80
Participants
  Day 3 | 54 | 55 | 15
  Week 1 | 54 | 58 | 32
  Week 2 | 59 | 53 | 38

8. Secondary Outcome: Change From Baseline in the Pruritus/Itch Score Reported in Participant Diaries at Day 3, Week 1 and Week 2
Description: Participants assessed the severity of their pruritus/itch during the daytime and nighttime (0=asymptomatic to 4=severe). The sum of the daytime and nighttime pruritus/itch scores could range from 0 to 8, with a higher score indicating greater severity. The changes from Baseline in the sum of the daytime and nighttime scores at the Day 3, Week 1 and Week 2 clinic visits were calculated.
Time Frame: Baseline Visit and Day 3 Visit, Week 1 Visit, Week 2 Visit
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Desloratadine 5 mg | Desloratadine 10 mg | Placebo
Number analyzed (Participants) | 80 | 79 | 80
Score on a Scale
  Change from Baseline at Day 3 | -2.37 [-2.74 to -2.00] | -2.73 [-3.10 to -2.36] | -0.50 [-0.87 to -0.13]
  Change from Baseline at Week 1 | -2.53 [-2.91 to -2.15] | -2.85 [-3.24 to -2.47] | -1.27 [-1.65 to -0.88]
  Change from Baseline at Week 2 | -2.85 [-3.30 to -2.41] | -2.97 [-3.42 to -2.51] | -1.75 [-2.23 to -1.27]

9. Secondary Outcome: Change From Baseline in Pruritus/Itch on a Visual Analog Scale (VAS) Reported by Participants at Day 3, Week 1 and Week 2
Description: Participants assessed the degree of their pruritus/itching using a 100-mm visual analog scale (VAS) (0 mm=No itch to 100 mm=Worst imaginable itch), with a higher score indicating more severe itching. The changes from Baseline in participant-assessed pruritus/itch at the Day 3, Week 1 and Week 2 clinic visits were calculated.
Time Frame: Baseline Visit and Day 3 Visit, Week 1 Visit, Week 2 Visit
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Desloratadine 5 mg | Desloratadine 10 mg | Placebo
Number analyzed (Participants) | 80 | 79 | 80
Score on a Scale
  Change from Baseline at Day 3 | -35.94 [-41.91 to -29.97] | -39.60 [-45.61 to -33.60] | -5.22 [-11.19 to 0.75]
  Change from Baseline at Week 1 | -40.82 [-46.55 to -35.09] | -48.82 [-54.60 to -43.03] | -15.88 [-21.63 to -10.13]
  Change from Baseline at Week 2 | -45.86 [-51.96 to -39.75] | -45.01 [-51.17 to -38.84] | -25.24 [-31.52 to -18.97]

10. Secondary Outcome: Change From Baseline in the Rash Score Reported in Participant Diaries at Day 3, Week 1 and Week 2
Description: Participants assessed the severity of their rash (erythema: 0=no symptom to 3=intensive redness, and wheal: 0=no symptom to 3=significant ridge). The sum score for erythema plus wheal could range from 0 to 6, with a higher score indicating greater severity. The changes from Baseline in the sum score for erythema plus wheal at the Day 3, Week 1 and Week 2 clinic visits were calculated.
Time Frame: Baseline Visit and Day 3 Visit, Week 1 Visit, Week 2 Visit
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Desloratadine 5 mg | Desloratadine 10 mg | Placebo
Number analyzed (Participants) | 80 | 79 | 80
Score on a Scale
  Change from Baseline at Day 3 | -2.21 [-2.57 to -1.85] | -2.31 [-2.67 to -1.94] | -0.77 [-1.13 to -0.40]
  Change from Baseline at Week 1 | -2.15 [-2.50 to -1.81] | -2.43 [-2.77 to -2.08] | -1.17 [-1.52 to -0.83]
  Change from Baseline at Week 2 | -2.51 [-2.88 to -2.13] | -2.45 [-2.83 to -2.06] | -1.70 [-2.11 to -1.29]

11. Secondary Outcome: Change From Baseline in the Dermatology Life Quality Index (DLQI) Total Score Reported by Participants at Week 1 and Week 2
Description: The DLQI is a 10-item questionnaire that measures how much participant skin problems have affected their life. Responses to questions about the effect of participant skin problems on life ranged from 0=Not at all to 3=Very much. The DLQI is broken down into 6 subscales: Symptoms and feelings (range 0-6), Daily activities (range 0-6), Leisure (range 0-6), Work and school (range 0-3), Personal relationships (range 0-6), and Treatment (range 0-3). DLQI subscales were summed to yield the DLQI total score, which could range from 0 to 30. For both DLQI subscales and DLQI total score, a higher score indicated a greater negative impact on life. Participants >=16 years of age completed the DLQI questionnaire about the condition of their skin over the previous week. The changes from Baseline in the DLQI total score at the Week 1 and Week 2 clinic visits were calculated.
Time Frame: Baseline Visit and Week 1 Visit, Week 2 Visit
Population: The FAS population consisted of all randomized participants who took at least one dose of study drug, had a Baseline assessment and at least one post-Baseline assessment for DLQI
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Desloratadine 5 mg | Desloratadine 10 mg | Placebo
Number analyzed (Participants) | 79 | 77 | 77
Score on a Scale
  Change from Baseline at Week 1 | -3.82 [-4.52 to -3.12] | -4.08 [-4.78 to -3.37] | -1.60 [-2.31 to -0.89]
  Change from Baseline at Week 2 | -4.10 [-4.83 to -3.38] | -4.01 [-4.74 to -3.28] | -2.53 [-3.28 to -1.78]

ADVERSE EVENTS:
Time Frame: Up to 4 weeks (Up to 2 weeks after last dose of study drug)
Description: The Safety Population consisted of all participants who received at least one dose of study drug. One Placebo group participant took the wrong study drug. This participant was analyzed separately.
Arm/Group | Desloratadine 5 mg | Desloratadine 10 mg | Placebo | Desloratadine 5 mg→Placebo
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/79 | 0/79 | 0/1
Other Adverse Events (participants affected / at risk) | 10/80 | 8/79 | 5/79 | 0/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Desloratadine 5 mg (N=80) | Desloratadine 10 mg (N=79) | Placebo (N=79) | Desloratadine 5 mg→Placebo (N=1)
Nasopharyngitis (Infections and infestations) | 8 (8) | 3 (3) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 3 (3) | 5 (6) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.